CLINICAL TRIAL: NCT04925362
Title: Identification of Clinical and Biological Factors Determining Disease Severity and Disease Progression in NAFLD: "THE FRENCH NATIONAL NAFLD COHORT" FRAMES (FRench pAtients With MEtabolic Steatosis)
Brief Title: THE FRENCH NATIONAL NAFLD COHORT (FRench pAtients With MEtabolic Steatosis)
Acronym: FRAMES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP190417; 2019-A01308-49 (Other: ANSM)
Record Dates: First submitted 2021-02-24; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: NAFLD; NASH; NASH - Nonalcoholic Steatohepatitis; Fibrosis; Cirrhosis
Keywords: Cohort
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Other): Patients with histologically confirmed NAFLD
  Interventions: Other: Biological specimens; Other: Additional visit

INTERVENTIONS:
Other: Biological specimens — Biological specimens are collected to better characterize patients of different severity and improve our understanding of clinical and histological heterogeneity at diagnosis :
  * added for the research : blood, urine, stools
  * collected for the research : liver tissue sample, if a liver biopsy is indicated for clinical reasons (standard of care)
Other: Additional visit — Visits if possible during standard care, otherwise added by the research (If necessary the annual visit will be added by research for the collection of biological samples)

SUMMARY:
The main objective of this cohort study is to determine genetic, clinical biologic and metabolic factors associated with patient heterogeneity in regards to severity of NAFLD at diagnosis as well as during the clinical course.

* at diagnosis, with the aim to better characterize patients of different severity and improve our understanding of clinical and histological heterogeneity at diagnosis
* during the clinical course to better understand and predict disease progression in terms notably of fibrosis progression and progression to cirrhosis

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is considered the hepatic manifestation of metabolic syndrome and is currently the most common cause of liver disease in many developed countries worldwide.

The aim of the study is to improve the scientific knowledge on markers associated with disease severity and progression in NAFLD.

The study is a multicentre French NAFLD cohort of well-characterized patients with biological samples covering the entire spectrum of NAFLD severity (steatosis, NASH, significant fibrosis, cirrhosis, hepatocellular carcinoma).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients with a confirmed diagnosis of NAFLD
3. Patients affiliated to French social security
4. Written informed consent signed by the patient

Exclusion Criteria:

1. Refusal or inability (lack of capacity) to give informed consent.
2. Average alcohol ingestion greater than 21/14 units/week (males/females) in the preceding 6 months or history of sustained excessive consumption of alcohol in past 5 years.
3. History or presence of Type 1 diabetes mellitus.
4. Presence of any other form of chronic liver disease except NAFLD
5. Recent (within 12 months) or concomitant use of agents known to cause hepatic steatosis (long-term systemic corticosteroids [>10 days], amiodarone, methotrexate, tamoxifen, tetracycline, high dose oestrogens, valproic acid).
6. Any contra-indication to liver biopsy.
7. Recent (within 3 months) change in dose/regimen or introduction of Vitamin E (at a dose ≥400 IU/day), betaine, s-adenosyl methionine, ursodeoxycholic acid, silymarin or pentoxifylline.
8. Non-French speaking/unable to access an interpreter.
9. Patients judged by the investigator to be unsuitable for inclusion in the study (e.g. judged by the physician as unlikely to be compliant with the study protocol).
10. Pregnant or breastfeeding women
11. Patient under legal protection measure (tutorship or curatorship) and patient deprived of freedom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2036-06 (Estimated); Study Completion 2036-06 (Estimated)

PRIMARY OUTCOMES:
Disease severity | Change of the fibrosis stage from baseline to 10 years
  The disease severity defined by the fibrosis stage on liver biopsy according to the semi-quantitative histological classification of NASH CRN.

SECONDARY OUTCOMES:
Ballooning grade | At baseline
Lobular inflammation | At baseline
  Composite scores of Lobular inflammation (Ballooning and Inflammation)
Steatohepatitis | At baseline
  Presence or Absence
Cirrhosis | Through study completion, an average of 10 years
  Cirrhosis defined by either :
  1. stage 4 of histological classification of fibrosis on liver biopsy or
  2. liver stiffness >14 kPa by elastometry
Obesity | Change from baseline to 10 years
  Obesity defined by either :
  1. Increased waist circumference by ethnically adjusted criteria or
  2. BMI ≥25
Type 2 diabetes | Change from baseline to 10 years
  Type 2 diabetes defined by Fasting glucose ≥100 mg/dL [5.6 mmol/L], HbA1c ≥48mmol/mol (6.5%) or previously diagnosed insulin resistance/type 2 diabetes mellitus (or on treatment).
Dyslipidaemia | Change from baseline to 10 years
  Dyslipidaemia defined by fasting TG level ≥150 mg/dL [1.7mmol/L]; or fasting HDL <40 mg/dL [1.03 mmol/L] in males and <50 mg/dL [1.29 mmol/L] in females; or on treatment);
Cardiovascular disease | Change from baseline to 10 years
  Cardiovascular disease defined by arterial hypertension (systolic BP ≥130 or diastolic BP ≥85 mmHg, or on antihypertensive treatment).
Necroinflammation measured by the activities component of the SAF | Change from baseline to 10 years
  Necroinflammation measured by the activities component of the SAF classification : ranges 0 to 4
  SAF : steatosis, activity, fibrosis
Necroinflammation measured by the NAS score | Change from baseline to 10 years
  Necroinflammation measured by the NAS score : ranges from 0 to 8
  NAS score : NAFLD Activity Score
Fasting insulin | Change from baseline to 10 years
Insulin sensitivity | Change from baseline to 10 years
  HOMA - %s

CONTACTS AND LOCATIONS:
Overall Officials: Vlad RATZIU, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No